CLINICAL TRIAL: NCT01644903
Title: Proteogenomic Monitoring and Assessment of Liver Transplant Recipients
Acronym: "Mini-Liver"
Status: Recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: The Scripps Research Institute (Other)
Responsible Party: Principal Investigator, Amna Daud, Transplant Hepatologist, Northwestern University
Other Study IDs: STU 26737
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Liver Transplant; Hepatitis C; Chronic Kidney Disease; Acute Rejection
MeSH Terms: conditions — Hepatitis C; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine Sample - One half cup of urine (100 mL) will be taken for research tests at each study visit.
  Blood Sample - About 1.5 tablespoons (20.5 mL) will be taken for research tests at each study visit.
  Liver Biopsy - A liver biopsy is a procedure to remove and examine a small piece of liver tissue. For this study, an extra tissue sample will possibly be taken during your biopsy. One additional needle pass may be made to collect the sample for this study.
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is being done to test blood, urine and tissue samples to see if this can help decide if CKD (Chronic Kidney Disease), AR (Acute Rejection) and HCV (Hepatitis C Virus) can be identified in its early stages. CKD damage to the kidneys, AR and HCV all lower the body's ability to function properly. Early detection of these conditions could assist with successful treatment and possibly lead to less repeat organ transplants.

DETAILED DESCRIPTION:
With the advent of more sensitive molecular techniques, biomarkers of kidney transplant rejection have been proposed that are potentially much more sensitive, specific and rapidly testable than conventional predictors of graft function such as GFR or tissue biopsies. Some of the early biomarkers during this evolution were the Cytotoxic T-cell (CTL) transcripts like perforin, granzyme B and fas ligand 11-13 for acute rejection. In the case of CAN/IFTA and CKD the molecular mechanisms and testable biomarkers also remain unclear. A few studies have reported the involvement of TGF-beta, extracellular matrix proteins like fibronectin and thrombopondin and tissue inhibitors of metalloproteins (TIMPs) as being upregulated in patients with Chronic Allograft Nephropathy (CAN/IFTA). Most of these studies were done in kidney transplant biopsies and the challenge of testing their expression and correlation in PBL as a minimally invasive tool was only addressed in a few studies. Another limitation of these first studies was the lack of the power to profile genes globally. To this end the advent of DNA microarrays has brought about a quantum leap in the ability to profile thousands of genes simultaneously. Thus far, microarray analysis has been reported in kidney transplant studies implicating gene signatures for acute rejection in transplant biopsies as well as for the first time by us in peripheral blood. To our knowledge only two studies have tried to profile CAN/IFTA in peripheral blood. A recent study attempted to validate three genes that were derived from a microarray analysis of kidney biopsies using RT-qPCR. All three genes were significantly differentially expressed in urine but not in PBL. Another study using microarrays showed that among a panel of 49 peripheral blood genes that were purported to distinguish "operational tolerance" in kidney rejection, 33 genes could also distinguish "chronic rejection" with 86% specificity.

Most of the studies in the literature, including our own, as well as our more recent unpublished peripheral blood gene expression studies of AR and CAN/IFTA reveal clear molecular signatures for both these forms of transplant outcomes. In sum, these data establish a first proof of concept that peripheral blood gene expression profiling can be used to develop markers of kidney allograft rejection and chronic kidney injury.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female recipients of all races, ≥18 years of age.
2. Patients undergoing primary or subsequent living or deceased donor liver transplantation.
3. Subject and/or guardian must be able to provide informed consent.
4. Subject and/or guardian must be able to comply with the study protocol.

Exclusion Criteria:

1. Inability or unwillingness of a participant and/or guardian to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The intention of our biomarker panel is to be broadly applicable to all patients with liver transplant with the assumption that there are common underlying molecular mechanisms of CKD and AR (and HCV) that can be detected hopefully at early stages of disease. We therefore want to validate and test our biomarker panel in a broad collection of patient types.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2010-04; Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Proteogenomic Biomarkers for CKD, AR and HCV | At time of liver biopsy
  To validate specific proteogenomic biomarker panels for CKD and AR (and HCV) in a prospective serial blood and urine monitoring study of liver transplant recipients

CONTACTS AND LOCATIONS:
Overall Officials: Josh Levitsky, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States